CLINICAL TRIAL: NCT02463045
Title: A Phase I Study to Evaluate the Safety/Tolerability and Pharmacokinetics of TOP1288 Rectal Single and Multiple Ascending Doses in Healthy Subjects and Multiple Doses in Subjects With Ulcerative Colitis
Brief Title: Study for Safety and Tolerability of TOP1288 Administered Rectally in Healthy and Ulcerative Colitis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Topivert Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TV-01
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2016-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (10):
- TOP1288 1mg (or placebo) (Experimental): TOP1288 1mg single dose or placebo
  Interventions: Drug: TOP1288
- TOP1288 10mg (or placebo) (Experimental): TOP1288 10mg single dose or placebo
  Interventions: Drug: TOP1288
- TOP1288 100mg (or placebo) (Experimental): TOP1288 100mg single dose or placebo
  Interventions: Drug: TOP1288
- TOP1288 200mg single dose or placebo (Experimental): TOP1288 200mg single dose or placebo
  Interventions: Drug: TOP1288
- TOP1288 400mg dose or placebo (Experimental): TOP1288 400mg (200mg bid) dose or placebo
  Interventions: Drug: TOP1288
- TOP1288 A mg or placebo (Experimental): TOP1288 A mg daily for 4 days
  Interventions: Drug: TOP1288
- TOP1288 B mg or placebo (Experimental): TOP1288 B mg daily for 4 days
  Interventions: Drug: TOP1288
- TOP1288 C mg or placebo (Experimental): TOP1288 C mg daily for 4 days
  Interventions: Drug: TOP1288
- TOP1288 D mg or placebo (Experimental): TOP1288 D mg bid for 4 days
  Interventions: Drug: TOP1288
- TOP1288 Xmg or placebo (Experimental): TOP1288 X mg od or bid for 4 days
  Interventions: Drug: TOP1288

INTERVENTIONS:
Drug: TOP1288
  Other Names: TOP1288 Placebo

SUMMARY:
This study evaluates the safety and tolerability of TOP1288 rectal single and multiple ascending doses in healthy subjects and multiple doses in subjects with ulcerative colitis.

DETAILED DESCRIPTION:
TOP1288, a narrow spectrum protein kinase inhibitor, is being developed as a novel, non-absorbed treatment for ulcerative colitis (UC). UC is a disease of unknown cause characterised by inflammation of the lining of the large intestine and manifesting with abdominal pain and bloody diarrhoea. TOP1288 given rectally has a local anti-inflammatory action in experimental models of UC. The present study will be the first time TOP1288 has been given to humans and explores the safety, tolerability and how the body handles (absorbs, distributes and eliminates) TOP1288 and seeks evidence of the biochemical effect of the drug in the body. The study is in three parts: Part 1 investigates single doses in groups of healthy volunteers, each group dosed with an increased dose provided the drug was safe and well tolerated at the previous level. Part 2 investigates multiple ascending doses in healthy volunteers each group dosed with an increased dose provided the drug was safe and well tolerated at the previous level. Part 3 investigates one dose level by administering that dose in patient volunteers with UC. The study design is adaptive - that is after the first dose level in Part 1, which is predefined, the exact dose and dose-intervals can be modified from a pre-set plan by a Safety Review Committee in the light of the emerging results.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects and Ulcerative Colitis Subjects

* Male or Female aged between 18 and 55 years (inclusive)
* Female subjects negative serum pregnancy test at Screening, non child-bearing potential.
* Body Mass Index between 18.0 and 29.9 kg/m2
* Good physical and mental health (other than ulcerative colitis for subjects in Part 3)
* Clinical laboratory test results within the reference ranges of the testing laboratory (with the exception of ulcerative colitis subjects with laboratory abnormalities consistent with their disease activity which will be allowed at Investigator's and the Sponsor's study physician/medical monitor's discretion)
* Blood pressure and pulse within normal range

Specific to Ulcerative Colitis Subjects

* Documented diagnosis of ulcerative colitis of at least 6 months duration confirmed by sigmoidoscopy
* Documented disease extending at least 15cm proximal from the anal verge
* Subject has experienced symptoms of ulcerative colitis on oral 5-ASA therapy in the 14 days before Screening and has been on stable dose regimen (no more than 2.4g/day) for at least 4 weeks duration prior to Day 1 and is willing to continue on this regimen for the duration of the study

Exclusion Criteria:

Healthy Subjects and Ulcerative Colitis Subjects

* Participation in another study of investigational medication within the last 3 months or 5 half-lives of the investigational medication, whichever is longer
* Positive for HIV 1/2 antibodies, hepatitis B surface antigen or hepatitis C antibodies
* Any prescription or non-prescription medications within prior 14 days (other than ulcerative colitis for subjects in Part 3 for whom a stable dose regimen of oral 5-ASA (no more than 2.4g/day) for at least 4 weeks before Day 1 is allowed and required)
* Consumption of any products containing caffeine or xanthine-related substances, foods or beverages containing Seville-type oranges or poppy seeds within 72 hours prior to admission
* Any acute or chronic illness (other than ulcerative colitis in Part 3) affecting the colon and/or rectum and/or anus, including haemorrhoids and irritable bowel syndrome, sufficient to cause symptoms and/or that in the judgement of the Investigator and the Sponsor's study physician/medical monitor would interfere with the subject's participation in the study
* Cardiovascular or cerebrovascular disease, including hypertension, angina, ischemic heart disease, transient ischaemic attacks, stroke and peripheral arterial disease sufficient to cause symptoms and/or require therapy to maintain stable status
* Abnormalities in haematology or ECG.
* Renal or liver impairment
* Active neoplastic disease or history of neoplastic disease within 5 years before Screening

Specific to Ulcerative Colitis Subjects

* Documented history of ulcerative colitis in immediate need of dose escalation of maintenance 5-aminosalicylate therapy.
* Proctitis at baseline endoscopy (on Day 1).
* Started oral 5-aminosalicylate within 4 weeks prior to baseline endoscopy or is not yet on a stable dose.
* Any medication administered per rectum within 1 week prior to baseline endoscopy.
* Oral or parenteral steroid within 2 weeks before the baseline endoscopy.
* Systemic immunomodulatory therapy (with the exception of azathioprine or 6-mercaptopurine in a dose regimen that is deemed acceptable for participation in the judgement of the Principal Investigator) within 12 weeks prior to baseline endoscopy.
* Previous treatment with biologic agents (including anti-TNF agents and vedolizumab) prior to baseline endoscopy.
* Mayo Score Physician's global assessment of 3, i.e., severe disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse events | To 7 days after the last dose
Safety as measured by clinical laboratory tests | To 7 days after the last dose
Safety as measured by vital signs | To 7 days after the last dose
Safety as measured by ECGs | To 7 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics profile single dose (AUC(0-24)); (Cmax); time to Cmax (tmax); apparent clearance (CL/F); apparent volume of distribution (Vz/F); mean residence time (MRT); elimination half-life (t½); elimination rate constant (λz) | To 72 hours post dose
  Single-dose PK (Day 1 Part 1, Part 2 and Part 3): Area under the concentration-time curve (AUC) from zero extrapolated to infinity (AUC(0-inf)); AUC from zero to the time of the last quantifiable concentration (AUC(0-t)); AUC from zero to the time of 12 hours (AUC(0-12)); AUC from zero to the time of 24 hours (AUC(0-24)); observed maximum concentration (Cmax); time to Cmax (tmax); apparent clearance (CL/F); apparent volume of distribution (Vz/F); mean residence time (MRT); elimination half-life (t½); elimination rate constant (λz).
Pharmacokinetics profile multiple dose AUC(0-t); (Ctrough); (Cmax,ss); (tmax,ss); (CLss/F); (Vz,ss/F); t½; λz; MRT; (0-tau) (RAUC); (RCmax); | To 72 hours post dose
  Multiple-dose PK (Day 4 in Part 2 and Part 3): AUC(0-t); AUC during the dosing interval (AUC(0-tau)); predose concentration (Ctrough); observed maximum concentration after multiple dosing (Cmax,ss); time to Cmax,ss (tmax,ss); apparent clearance at steady state (CLss/F); apparent volume of distribution at steady state (Vz,ss/F); t½; λz; MRT; accumulation ratio for AUC(0-tau) (RAUC); accumulation ratio for Cmax (RCmax); time independency factor.

CONTACTS AND LOCATIONS:
Locations (1):
- CTU, London, United Kingdom